CLINICAL TRIAL: NCT03720743
Title: Effect of a Biodanza Program on Desire, Excitation and Sexual Inhibition in Young Adults. A Randomized Pilot Study
Brief Title: Effect of Biodanza on Desire, Excitation and Sexual Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, María del Mar Lopez-Rodriguez, Assistant Professor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: amuelle
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sexual Desire Disorder; Sexual Arousal Disorder; Sexual Inhibition
Keywords: Biodanza; libido; sexual excitement; sexual inhibition; young adults; dance therapy; complementary therapies
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodanza (Experimental): Intervention group received a total of 10 sessions, once a week, over the course of two months. Each session lasted 60 minutes. All sessions began with a 10-minute warm-up period combining music and low-intensity movements as a welcome round, followed individual exercises, in pairs and/or groups, which included dance combined with exercises based on the five lines of Biodanza (vitality, sexuality, creativity, affectivity and transcendence). Finally, a celebration and farewell round of 10 minutes was held. At the end of each session, the participants were asked to share their experiences with the rest of the group.
  Interventions: Other: Biodanza
- Control Group (No Intervention): The study allowed control group subjects to participate in Biodanza sessions after the follow-up period.

INTERVENTIONS:
Other: Biodanza — Intervention group received a total of 10 sessions, once a week, over the course of two months. Each session lasted 60 minutes. All sessions began with a 10-minute warm-up period combining music and low-intensity movements as a welcome round, followed individual exercises, in pairs and/or groups, which included dance combined with exercises based on the five lines of Biodanza (vitality, sexuality, creativity, affectivity and transcendence). Finally, a celebration and farewell round of 10 minutes was held. At the end of each session, the participants were asked to share their experiences with the rest of the group.
  Other Names: Dance
  Arms: Biodanza

SUMMARY:
the objective of this study was to examine the effects of a 10 weeks biodanza program on the sexual desire and inhibition/arousal of a sample of healthy young adults.

A randomized clinical study was carried out, involving a total of 86 young adults divided into Intervention Group (BG) and Control Group (CG), carrying out biodanza sessions during 10 weeks. The Sexual Desire Inventory (SDI) and the Sexual Inhibition/Sexual Arousal-Short Form Scale (SIS/SES-SF) were completed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* having correctly completed the online questionnaire.
* to attend a minimum of eight Biodanza sessions.

Exclusion Criteria:

* exceed 30 years old.
* the presence of some type of physical or mental disability that could prevent their participation in the therapy or the completion of the questionnaires.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Sexual desire | 3 months
  Sexual Desire Inventory (SDI) formed by 13 items, divided into dyadic sexual desire (Dyadic SD) (items 1-9) and solitary sexual desire (Solitary SD) (items 10-13), and valued by a Likert scale according to frequency (0 = never, and 7 = more than once a day), and intensity (0 = not desire, and 8 = strong desire), in a total range between 0 and 101 points, being higher the desire the greater the response result.
Sexual excitement/sexual inhibition | 3 months
  Sexual Inhibition/Sexual Excitement Scales - Short Form consists of 14 items with responses assessed using a Likert scale 1-4 (1 = completely agree; 4 = completely disagree) that measure three sub-scales: Sexual Excitation Scale (SES) (items 1, 3, 8, 10, 11, 14) with a score range between 4 and 16; Sexual Inhibition Scale 1 (SIS1) (items 4, 9, 12, 13) related to distraction/concentration in sexual performance, with a range between 4 and 16, and Sexual Inhibition Scale 2 (SIS2) (items 2, 5, 6, 7) related to the fear to be discovered or to contract some type of sexually transmitted infection (STI), with a range between 4 and 16.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No